CLINICAL TRIAL: NCT03413618
Title: The Efficacy of Rivaroxaban With Diosmin in the Long-term Treatment of Acute Proximal Deep Vein Thrombosis
Brief Title: Rivaroxaban With Diosmin in Long-term Treatment of Deep Vein Thrombosis
Acronym: RIDILOTT-DVT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIDILOTT-DVT
Record Dates: First submitted 2018-01-18; First posted 2018-01-29 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2019-07

CONDITIONS: Deep Vein Thrombosis; Postthrombotic Syndrome
Keywords: deep vein thrombosis; postthrombotic syndrome; anticoagulation; treatment; prevention
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome | interventions — Rivaroxaban; Diosmin; Stockings, Compression

STUDY DESIGN:
Intervention Model Description: Randomized open-labeled clinical trial with a masked outcomes assessor
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor does not involve in randomisation and treatment process, has no information about the patient's belonging to one of the study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Rivaroxaban + Diosmin + Stockings (Experimental): treatment of deep vein thrombosis with anticoagulation (rivaroxaban), elastic compression stockings and additional prescription of diosmin
  Interventions: Drug: Rivaroxaban; Drug: Diosmin; Other: compression stockings
- Control: Rivaroxaban + Stockings only (Active Comparator): standard treatment of deep vein thrombosis with anticoagulation (rivaroxaban) and elastic compression stockings
  Interventions: Drug: Rivaroxaban; Other: compression stockings

INTERVENTIONS:
Drug: Rivaroxaban — 15 mg b.i.d. for 3 weeks and then 20 mg q.d. up to 6 month
  Other Names: xarelto
Drug: Diosmin — 600 mg q.d. for 12 month
  Other Names: flebodia
  Arms: Experimental: Rivaroxaban + Diosmin + Stockings
Other: compression stockings — above knee stocking for 12 month

SUMMARY:
The randomized clinical study aimed to assess the efficacy and safety of standard anticoagulation with rivaroxaban in combination with diosmin compared to the isolated use of standard rivaroxaban for prolonged therapy of acute femoro-popliteal deep vein thrombosis reflected the speed of deep vein recanalization and incidence of post-thrombotic syndrome.

DETAILED DESCRIPTION:
Deep vein thrombosis is an acute inflammatory disease that affects vein wall and leads to the structural changes in the wall and valves reflected with chronic venous insufficiency that called postthrombotic syndrome (PTS).

Diosmin as a flavonoid agent has properties to reduce leukocyte-endothelial interaction and inflammatory response, that could reduce the damage to venous wall and valves.

The hypothesis of the study is based on assumption that diosmin combined with standard anticoagulation can improve outcomes of femoro-popliteal DVT due to increase speed of veins recanalization, decrease of vein wall inflammation and finally decrease the incidence of PTS at 6 month and 1 year after index DVT.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* The first episode of femoro-popliteal deep vein thrombosis (DVT)
* Verification of DVT by duplex ultrasound
* Informed consent signed

Exclusion Criteria:

* Suspicion of pulmonary embolism (PE)
* Verified PE
* Bilateral DVT
* Contraindications for rivaroxaban (in accordance with the official instructions)
* Contraindications for diosmin (in accordance with the official instructions)
* Active cancer
* Verified severe thrombophilia (antiphospholipid antibodies, deficiency of proteins C, S, antithrombin 3)
* Use of other anticoagulants for more than 7 days from the DVT verification
* Impossibility of using compression stocking after 3 days from DVT verification
* Performed surgical intervention on the superficial or deep veins of the lower extremities (thrombolysis, thrombectomy, vein ligation, implantation of the inferior cava filter)
* Continuous use of other drugs that affect the hemostasis system (except for acetylsalicylic acid in a dose of not more than 100 mg).
* Low compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Schastlivtsev, PhD, Principal Investigator — Pirogov Russian National Research Medical University
Locations (1):
- Clinical Hospital no.1 of the President's Administration of Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lobastov K, Sautina E, Alencheva E, Bargandzhiya A, Schastlivtsev I, Barinov V, Laberko L, Rodoman G, Boyarintsev V. Intermittent Pneumatic Compression in Addition to Standard Prophylaxis of Postoperative Venous Thromboembolism in Extremely High-risk Patients (IPC SUPER): A Randomized Controlled Trial. Ann Surg. 2021 Jul 1;274(1):63-69. doi: 10.1097/SLA.0000000000004556. PMID 33201130

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Admitted to the hospital with the suspicion for DVT: 202; DVT verified: 158; Eligible DVT: 102; Rejected to participate: 12; Randomized: 90
Groups:
- Experimental: Rivaroxaban + Diosmin + Stockings: treatment of DVT with anticoagulation (rivaroxaban), elastic compression stockings and additional prescription of diosmin
  Rivaroxaban: 15 mg b.i.d. for 3 weeks and then 20 mg q.d. up to 6 month
  Diosmin: 600 mg q.d. for 12 month
  compression stockings: above knee stocking for 12 month
- Control: Rivaroxaban + Stockings Only: standard treatment of DVT with anticoagulation (rivaroxaban) and elastic compression stockings
  Rivaroxaban: 15 mg b.i.d. for 3 weeks and then 20 mg q.d. up to 6 month
  compression stockings: above knee stocking for 12 month
Period: Overall Study
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stockings | Control: Rivaroxaban + Stockings Only
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Rivaroxaban + Diosmin + Stocking: treatment of DVT with anticoagulation (rivaroxaban), elastic compression stockings and additional prescription of diosmin
  Rivaroxaban: 15 mg b.i.d. for 3 weeks and then 20 mg q.d. up to 6 month
  Diosmin: 600 mg q.d. for 12 month
  compression stockings: above knee stocking for 12 month
- Total: Total of all reporting groups
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stocking | Control: Rivaroxaban + Stockings Only | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (13.8) | 60.2 (13.1) | 58.8 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 28 | 28 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 45 | 45 | 90
Time to randomization [Mean (Standard Deviation); unit: days] — Number of days from DVT verification to randomization
  days | 3.4 (1.2) | 3.5 (1.6) | 3.5 (1.4)
Unprovoked DVT [Count of Participants; unit: Participants] — DVT without any identified clinical provocation (e.g. major surgery, trauma, immobilization, pregnancy and postpartum, estrogen-containing pills, long-travel, etc)
  Participants | 29 | 33 | 62
Preexisting chronic venous disease [Count of Participants; unit: Participants] — Chronic venous disease (CVD) according to the Clinical-Etiology-Anatomy-Pathophysiology (CEAP) clinical class: C0 - no signs for CVD; C1 - telangiectasia and reticular veins; C2 - varicose veins; C3 - venous edema; C4 - skin pigmentation, induration, venous eczema of skin white atrophy; C5 - healed venous ulcer; C6 - active venous ulcer. Preexisting CVD suggests C2 and higher CEAP clinical class.
  Participants | 23 | 32 | 55
Thrombus burden [Mean (Standard Deviation); unit: Marder score] — Extension of DVT assessed with duplex ultrasound by Marder score (see Appendix 1 to the Protocol): ranges from 0 (no thrombus) to 34 (occlusion of all veins in one limb).
  Marder score | 15.2 (4.7) | 11.6 (4.1) | 13.4 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postthrombotic Syndrome as Determined by Villalta Score
Description: Detection of the postthrombotic syndrome (PTS) was made according to the Villalta score (a combination of 5 subjective symptoms and 6 objective signs of chronic venous disease) ranged from 0 (no signs) to 33 scores (maximal severity). PTS defined as 5 and more scores; mild PTS as 5-9 scores; moderate PTS as 10-14 scores; severe PTS as 15 and more scores.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stockings | Control: Rivaroxaban + Stockings Only
Number analyzed (Participants) | 45 | 45
Participants | 3 | 22
Statistical Analysis 1: Comparison: Experimental: Rivaroxaban + Diosmin + Stockings vs Control: Rivaroxaban + Stockings Only; Test type: Superiority; p < 0.0001, Fisher Exact

2. Secondary Outcome: Number of Participants With Recurrent Symptomatic or Asymptomatic DVT
Description: detection of any episode of recurrent DVT with or without clinical signs verified by duplex ultrasound
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stockings | Control: Rivaroxaban + Stockings Only
Number analyzed (Participants) | 45 | 45
Participants | 1 | 6
Statistical Analysis 1: Comparison: Experimental: Rivaroxaban + Diosmin + Stockings vs Control: Rivaroxaban + Stockings Only; Test type: Superiority; p = 0.049, Log Rank

3. Secondary Outcome: Number of Participants With Symptomatic Pulmonary Embolism
Description: detection of symptomatic pulmonary embolism verified with CT pulmonary angiogram
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stockings | Control: Rivaroxaban + Stockings Only
Number analyzed (Participants) | 45 | 45
Participants | 0 | 0

4. Secondary Outcome: The Value of Venous Clinical Severity Score
Description: Venous Clinical Severity Score (VCSS) is a combination of subjective symptoms and objective signs of CVD aimed to assess the severity of disease and ranges from 0 (no signs and symptoms of CVD) to 30 (severe signs and symptoms of CVD)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: VCSS score
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stockings | Control: Rivaroxaban + Stockings Only
Number analyzed (Participants) | 45 | 45
VCSS score | 1.2 (1.1) | 4.4 (2.1)
Statistical Analysis 1: Comparison: Experimental: Rivaroxaban + Diosmin + Stockings vs Control: Rivaroxaban + Stockings Only; Test type: Superiority; p < 0.0001, Fisher Exact

5. Secondary Outcome: The Value of Chronic Lower Limb Venous Insufficiency Questionnaire - 20 Items
Description: Chronic Lower Limb Venous Insufficiency Questionnaire - 20 items (CIVIQ-20) is a venous specific questionnaire to assess the disease-specific quality of life (QoL). It contains 20 items of 1-5 scores, totally, from 20 (best QoL) to100 (worst QoL) scores.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: CIVIQ-20 scores
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stockings | Control: Rivaroxaban + Stockings Only
Number analyzed (Participants) | 45 | 45
CIVIQ-20 scores | 22.1 (3.3) | 28.8 (7.6)
Statistical Analysis 1: Comparison: Experimental: Rivaroxaban + Diosmin + Stockings vs Control: Rivaroxaban + Stockings Only; Test type: Superiority; p < 0.0001, Fisher Exact

6. Secondary Outcome: Number of Participants With Full Recanalization of the Popliteal Vein
Description: Full recanalization of popliteal vein suggests the residual venous obstruction (RVO) less than 20%. The RVO was assessed by duplex ultrasound and calculated as the vein cross-sectional diameter under the maximal compression divided on the diameter without any compression multiplied by 100%.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stockings | Control: Rivaroxaban + Stockings Only
Number analyzed (Participants) | 45 | 45
Participants | 42 | 28

7. Secondary Outcome: Extension of Residual Venous Obstruction by Marder Score
Description: Residual venous obstruction (RVO) defined as a thrombotic masses occupying 20% and more of the vein cross-sectional diameter was measured by duplex ultrasound and calculated as the vein cross-sectional diameter under the maximal compression divided on the diameter without compression and multiplied by 100%. The extension of RVO was assessed by Marder score, the sum of all affected venous segments, evaluated by different scores (see Appendix of the Protocol), that ranged from 0 (no RVO) to 34 (RVO in all possible venous segments in one limb).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Marder score
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stockings | Control: Rivaroxaban + Stockings Only
Number analyzed (Participants) | 45 | 45
Marder score | 0.3 (1.0) | 1.9 (2.4)
Statistical Analysis 1: Comparison: Experimental: Rivaroxaban + Diosmin + Stockings vs Control: Rivaroxaban + Stockings Only; Test type: Superiority; p = 0.001, Fisher Exact

8. Secondary Outcome: Adverse Events
Description: any adverse events detected or suspected
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stockings | Control: Rivaroxaban + Stockings Only
Number analyzed (Participants) | 45 | 45
Participants | 5 | 4
Statistical Analysis 1: Comparison: Experimental: Rivaroxaban + Diosmin + Stockings vs Control: Rivaroxaban + Stockings Only; Test type: Superiority; p = 1.000, Fisher Exact

9. Secondary Outcome: Major Bleeding
Description: according to the International Society of Thrombosis and Hemostasis (ISTH) definition, major bleeding defined as fatal bleeding, and/or symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a fall in hemoglobin level of 20 g/L or 1.24 mmol/L or more, or leading to transfusion of two or more units of whole blood or red cells
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stockings | Control: Rivaroxaban + Stockings Only
Number analyzed (Participants) | 45 | 45
Participants | 0 | 0

10. Secondary Outcome: Clinically Relevant Non-major Bleeding
Description: any non-major bleeding requiring anticoagulant withdrawal, and/or performing haemostatic measures, and/or hospitalization, and/or an unscheduled medical appointment
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stockings | Control: Rivaroxaban + Stockings Only
Number analyzed (Participants) | 45 | 45
Participants | 1 | 2

11. Secondary Outcome: Minor Bleeding
Description: any non-major or non-clinically relevant bleeding does not require the suspension of therapy and changes in the patient's lifestyle
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Rivaroxaban + Diosmin + Stockings | Control: Rivaroxaban + Stockings Only
Number analyzed (Participants) | 45 | 45
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Study Group: treatment of DVT with anticoagulation (rivaroxaban), elastic compression stockings and additional prescription of diosmin
  Rivaroxaban: 15 mg b.i.d. for 3 weeks and then 20 mg q.d. up to 6 month
  Diosmin: 600 mg q.d. for 12 month
  compression stockings: above knee stocking for 12 month
- Control Group: standard treatment of DVT with anticoagulation (rivaroxaban) and elastic compression stockings
  Rivaroxaban: 15 mg b.i.d. for 3 weeks and then 20 mg q.d. up to 6 month
  compression stockings: above knee stocking for 12 month
Arm/Group | Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 5/45 | 4/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=45) | Control Group (N=45)
Dispesia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Clinically relevant non-major bleeding (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Minor bleeding (Blood and lymphatic system disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Unsuspected high frequency of PTS in the Control group (standard treatment with rivaroxaban and compression stockings) led to early termination of enrollment (75% of planned sample size).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT03413618/Prot_SAP_000.pdf